CLINICAL TRIAL: NCT07361783
Title: The Impact of Injection of a Loading Dose of Unfractionated Heparin on Patients With Acute ST-segment Elevation Myocardial Infarction Scheduled for Primary PCI at Initial Medical Contact: A Multicenter, Prospective, Randomized Controlled Study（HELP-PCI 2）
Brief Title: Impact of Pre-Hospital Heparin Loading in STEMI Patients for Primary PCI: The HELP-PCI 2 Trial
Acronym: HELP-PCI 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Jing (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Xianning Central Hospital (Other); Hubei University of Medicine (Other); Yichang Central People's Hospital (Other); Xiangyang Central Hospital (Other); Caidian District People's Hospital (Unknown); Chibi People's Hospital (Unknown); Jiangxia First People's Hospital (Unknown); Anlu Pu'ai Hospital (Unknown); Jingzhou Central Hospital (Other); The Fifth Hospital of Wuhan (Other); Shiyan People's Hospital (Unknown); The Third People's Hospital of Hubei Province (Other); China Resources Wugang General Hospital (Unknown); Wuhan Puren Hospital (Other); Sinopharm Dongfeng General Hospital (Unknown); Changjiang Shipping General Hospital (Unknown); Wuhan No.1 Hospital (Other); Wuhan No.3 Hospital (Unknown); Xishui County People's Hospital (Unknown); Xiangyang Hospital of Traditional Chinese Medicine (Unknown); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Jiangling People's Hospital (Unknown); Wuhan No.6 Hospital (Unknown); The Central Hospital of Huanggang (Other); Laohekou First Hospital (Unknown); Wuxue First People's Hospital (Unknown); Hanyang University (Other); The First People's Hospital of Tianmen (Unknown); Xianning First People's Hospital (Unknown); Wuhan Hospital of Traditional Chinese Medicine (Other); Wuhan Central Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Second Xiangya Hospital of Central South University (Other); Tongcheng People's Hospital of Anhui province (Unknown); Songzi People's Hospital (Unknown); Xiantao First People's Hospital (Unknown); Ezhou Central Hospital (Unknown); People's Hospital of Jingshan (Unknown)
Responsible Party: Sponsor-Investigator, Chen Jing, MD, PhD, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WDRM2025-K023
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Primary PCI; ST-elevation Myocardial Infarction (STEMI)
Keywords: Heparin; Primary Percutaneous Coronary Intervation; ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Heparin at the first medical contact (Experimental): The experimental group was treated with a loading dose of 100U/kg of unfractionated heparin at the first medical contact
  Interventions: Drug: Unfractionated heparin
- Administration of Heparin in the catheterization laboratory (Active Comparator): the control group was treated with a loading dose of 100U/kg of unfractionated heparin in the catheterization laboratory.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Unfractionated heparin — An intravenous injection of 100 U/kg of UFH will be given at first medical contact before primary PCI (if assigned to experimental group) or in the catheter lab through the arterial sheath when starting primary PCI (if assigned to control group)

SUMMARY:
This randomized, multicenter, prospective trial will enroll 6,294 participants in approximately 80 centers. STEMI patients with onset time within 12 hours and scheduled for primary PCI will be randomly assigned to two groups in a 1:1 ratio. Patients meeting the criteria were randomly assigned. It is recommended that loading doses of dual antiplatelet therapy be administered immediately after electrocardiogram diagnosis. The experimental group was required to be given an intravenous injection of 100 U/kg of UFH within 10 minutes after randomization, and this should be completed at least before delivery to the catheter lab. The control group was recommended to be given 100 U/kg of UFH through the arterial sheath, but the actual intraoperative dosage was determined by the interventional cardiologist. No patient is allowed to use low-molecular-weight heparin, bivalirudin, glycoprotein IIb/IIIa inhibitors or other antithrombotic drugs before coronary angiography. The planned enrollment period for this study is 24 months. The scheduled follow-up visits will occur at 30 days (±7 days), 3 months (±14 days), and if conditions permit, at 6 months (±30 days) and 1 year (±30 days) after randomization. The purpose of this study is to evaluate the composite endpoint of all-cause death, recurrent myocardial infarction, urgent coronary revascularization, stent thrombosis, or stroke within 30 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. STEMI within 12 hours of onset Newly developed adjacent two or more leads with ST segment elevation of ≥1mm (lead V2-V3 elevation of ≥2mm).

   Newly developed left bundle branch block (LBBB). In the right bundle-branch block (RBBB), the ST segment of leads V1-V3 is elevated or Q waves occur.
3. Primary PCI was planned if the time from first medical contact to balloon dilatation was expected to be less than 120 minutes.

Exclusion Criteria:

1. Thrombolytic therapy recipients;
2. Currently taking oral anticoagulant drugs or having been treated with heparin, low molecular weight heparin, suldaparinol sodium, bivalirudin or IIb/IIIa receptor antagonists within 48 hours before randomization;
3. Patients undergoing cardiopulmonary resuscitation;
4. Patients with cardiogenic shock;
5. Combined mechanical complications (rupture of the free wall of the heart, perforation of the ventricular septum, insufficiency or rupture of the papillary muscle leading to severe mitral regurgitation);
6. History of intracranial parenchymal aneurysm, intracranial arteriovenous malformation, intracranial hemorrhage, ischemic stroke or transient ischemic attack within the last 6 months, and active hemorrhage within the last 2 weeks;
7. Major surgery within one month;
8. Previous history of CABG;
9. Patients with a history of heparin-induced thrombocytopenia or those known to be allergic to anticoagulant or antiplatelet drugs;
10. Combined with other serious diseases and life expectancy less than 12 months;
11. Pregnant or lactating women;
12. Currently participating in clinical research on other drugs or devices;
13. Refuse to sign the informed consent form;
14. The researcher judged that it was not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6294 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
The composite endpoint of all-cause death, recurrent myocardial infarction, urgent coronary revascularization, stent thrombosis, or stroke within 30 days after randomization | Within 30 days after randomization.
  The composite endpoint of all-cause death, recurrent myocardial infarction, urgent coronary revascularization, stent thrombosis, or stroke within 30 days after randomization
Primary safety endpoint: Major bleeding (BARC type 3~5) within 30 days | within 30 days after randomization
  Major bleeding (BARC type 3~5)

SECONDARY OUTCOMES:
Net Clinical Adverse Event | With 30 days and 90 days after randomization
  Composite of all-cause death, recurrent myocardial infarction, urgent coronary revascularization, stent thrombosis, stroke, and BARC type 3-5 bleeding
Individual Clinical Adverse Event | Within 30 days and 90 days after randomization
  all-cause death, cardiovascular death, recurrent myocardial infarction, urgent coronary revascularization, stent thrombosis, or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, PhD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No